CLINICAL TRIAL: NCT02992483
Title: Phase I Open Label, Multi-center Study to Characterize the Safety, Tolerability and Pharmacokinetics of Intravenously Administered MIK665, a Mcl-1 Inhibitor, in Patients With Refractory or Relapsed Lymphoma or Multiple Myeloma
Brief Title: Phase I Study of MIK665, a Mcl-1 Inhibitor, in Patients With Refractory or Relapsed Lymphoma or Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMIK665X2101; 2016-003624-22 (EudraCT Number)
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Multiple Myeloma (MM), Lymphoma, Large B-Cell, Diffuse (DLBCL), Lymphoma
Keywords: multiple myeloma; lymphoma; dlbcl
MeSH Terms: conditions — Multiple Myeloma; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MIK665 (Experimental)
  Interventions: Drug: MIK665

INTERVENTIONS:
Drug: MIK665 — MIK665
  Other Names: S64315

SUMMARY:
The purpose of this first in human study is to assess safety, tolerability, PK and preliminary clinical activity and to estimate the MTD(s)/RDE(s) of MIK665 (also referred as S64315) as single agent administered intravenously (i.v.) in adult patients with refractory or relapsed lymphoma or multiple myeloma.

DETAILED DESCRIPTION:
The design of this phase I, open label, dose finding study was chosen in order to characterize the safety and tolerability of MIK665 and to determine the Maximal Tolerated Dose(s) (MTD(s)) and/or Recommended Dose(s) for Expansion (RDE(s)).

This study will utilize a Bayesian Hierarchical model to guide dose escalation and estimate the MTD(s) based on the dose-DLT relationship(s) for MIK665 in the indications.

The expansion part of the study will employ an open-label multiple arm design. The purpose of the expansion part is to further assess safety, tolerability, PK, PD and the anti-tumor activity of MIK665 at the selected RDE/s for Multiple Myeloma (MM) and MYC positive Diffuse large B-Cell Lymphoma (DLBCL) identified in the dose-escalation part.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years.
* Histologically confirmed lymphoma (WHO classification), or confirmed MM (IMWG), that is relapsed and/or refractory.
* Other Inclusion Criteria May Apply.

Exclusion Criteria

* Known history of chronic liver disease
* History of chronic pancreatitis.
* Prior treatment with Mcl-1 inhibitor.
* Other Exclusion Criteria May Apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of AEs and SAEs, incl. changes in laboratory parameters, vital signs and ECGs. | 2 years
Incidence of DLTs during the first cycle of treatment with single agent MIK665 during the dose escalation phase only | 2 years
Tolerability: Dose interruptions | 2 years
Tolerability: Dose reductions | 2 years
Tolerability: Dose intensity | 2 years

SECONDARY OUTCOMES:
Best Overall response (BOR) per International Myeloma Working Group (IMWG) criteria for Myeloma; and per revised criteria for staging of the International Working Group (IWG) guidelines for Lymphoma | 2 years
Area Under Curve (AUC) | 2 years
  Plasma PK parameter
Maximum Plasma Concentration (Cmax) | 2 years
  Plasma PK parameter
Terminal elimination half-life (T1/2) | 2 years
  Plasma PK parameter
Apparent volume of distribution (Vz) | 2 years
  Plasma PK parameter
Clearance (CL) | 2 years
  Plasma PK parameter
Duration of Response (DOR)per International Myeloma Working Group (IMWG) criteria for Myeloma; and per revised criteria for staging of the International Working Group (IWG) guidelines for Lymphoma | 2 years
Progression Free Survival (PFS) per International Myeloma Working Group (IMWG) criteria for Myeloma; and per revised criteria for staging of the International Working Group (IWG) guidelines for Lymphoma | 2 years

CONTACTS AND LOCATIONS:
Locations (8):
- MD Anderson Cancer Center/University of Texas MD Anderson CC, Houston, Texas, United States
- Novartis Investigative Site, Heidelberg, Victoria, Australia
- Novartis Investigative Site, Nantes, France
- Germany (2):
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Kiel
- Novartis Investigative Site, Rozzano, MI, Italy
- Novartis Investigative Site, Fukuoka, Fukuoka, Japan
- Novartis Investigative Site, Salamanca, Castille and León, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17854